CLINICAL TRIAL: NCT05104944
Title: A Randomised Feasibility Trial to Define Outcome Measures for Acute Charcot Neuroarthropathy in Diabetes and Their Use in Assessing Clinical Management (CADOM)
Brief Title: Defining Outcome Measures for Acute Charcot Neuroarthropathy in Diabetes and Their Use in Assessing Clinical Management
Acronym: CADOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Collaborators: University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 222668 (15-01-16); ICA-CDRF-2015-01-050 (Other Grant/Funding Number: NIHR)
Record Dates: First submitted 2021-04-29; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Diabetes
Keywords: Charcot neuroarthropathy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Intervention: Serial use of MRI at 3, 6, 9 and 12 months to identify disease resolution and thus discontinue immobilisation in addition to standard care
Masking Description: It is not possible to blind this study due to the nature of reporting the MRIs, whereby comparison is made with the previous images, which indicates the trial arm the participant has been randomised to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Intervention - Standard Care and Serial MRIs) (Experimental): Immobilisation discontinued on the basis of MRI defined disease resolution at 3, 6, 9 or 12 months. In the intervention arm participants will receive additional MRIs at 3, 6, 9 and 12 months. Patients randomised to serial MRI will not undergo further MRI once remission has been diagnosed i.e. if remission is diagnosed at 6 months the MRI at 9 and 12 months will not occur.
  Interventions: Radiation: Serial MRIs
- Arm B (Control - Standard Care and one additional MRI) (No Intervention): Immobilisation discontinued on the basis of clinical remission determined by skin temperature measurement and MRI. In the standard care arm participants will receive one additional MRI when the temperature measurements, X-ray and/or signs and symptoms indicate to the clinical team that the foot is in remission. A temperature difference of ≤ 2ºC which is maintained or improves on two separate consecutive occasions for a period of ≥4weeks will be the indicator to arrange the second MRI, to confirm the diagnosis of remission. If participants in either arm of the trial have not reached remission at the end of the 12 month active phase of the study they will exit the study. Ongoing standard care will be provided by their clinical team.

INTERVENTIONS:
Radiation: Serial MRIs — Serial use of MRI at 3, 6, 9 and 12 months to identify disease resolution and thus discontinuation of immobilisation plus standard care.
  Other Names: Serial use of MRI at 3, 6, 9 and 12 months
  Arms: Arm A (Intervention - Standard Care and Serial MRIs)

SUMMARY:
The aim of this study is to explore the use of serial magnetic resonance imaging (MRI) in an attempt to reduce the duration of immobilisation of the foot and thereby reduce the morbidity associated with its routine management and reduce costs. The project will have two components: a feasibility study and embedded within this a qualitative study of the patient's perspective of the experience of being diagnosed with Charcot neuroarthropathy (CN) and undergoing treatment.

DETAILED DESCRIPTION:
The aim of the study is to assess the feasibility of using serial magnetic resonance imaging (MRI) to reduce treatment times in Charcot in people with diabetes.

Charcot is a devastating complication for people who develop it. There are over 4000 new cases of Charcot diagnosed every year. If the inflammation goes on for long enough it can cause fractures and dislocations within the foot, which left untreated can lead to foot deformity and complications such as ulcerations.

A diagnosis of Charcot has been shown to reduce people's quality of life. People who have had this condition die on average 14years younger than the general population. Every year about 50-100 people who have been diagnosed with Charcot neuroarthropathy undergo an amputation of their leg.

Charcot is treated by wearing a non-removable cast or boot. No-one knows how long this treatment should last, some recommend 6 months, others more than a year. Early treatment has been shown to lead to fewer complications.

There is some information from small studies that repeated assessment with MRI may prove useful in helping clinicians decide when to stop treatment, and it may decrease treatment times.

This study will be a feasibility study involving 60 people. Patients will be recruited from hospital run Diabetic Foot Clinics. Patients will be randomised to either receive MRI at baseline 3,6,9 and 12 months or to receive current usual care; repeated foot temperature measurements and x-rays. If the study results indicate the study is feasible to do, the information will be used to design a much larger study.

Some patients will also be asked to participate in an interview at the end of the study, to gain insights into their experience of having Charcot and involvement in the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are willing and have capacity to give informed consent
* People with diabetes as diagnosed by the WHO criteria
* Age 18 years or over
* New or suspected diagnosis of acute CN (no previous incidence of acute CN within the last 6 months on the same foot) treated with off-loading
* Understand written and verbal instructions in English

Exclusion Criteria:

* People who have received a transplant and others receiving immunosuppressant therapy or using long term oral glucocorticoids other than in the routine management of glucocorticoid deficiency. Participants on a low doses of oral glucocorticoids (<10mgs for ≤7 days) are eligible to participate in the study.
* Participation in another intervention study on active CN
* Contra-indication for MRI
* Treatment for previous suspected CN on the same foot in the last 6 months
* Suspected or confirmed bilateral active CN at presentation
* Active osteomyelitis at randomisation
* Previous contralateral major amputation
* Inability to have an MRI scan
* Patients receiving palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who meet eligibility criteria. | through study completion, an average of 4 years
  Feasibility outcome.
The number of eligible patients recruited. | through study completion, an average of 4 years
  Feasibility outcome.
The number of participants in which an alternative diagnosis of the foot disease is made during the intervention phase of the trial. | through study completion, an average of 4 years
  Feasibility outcome.
The proportion of patients that withdraw or are lost to follow up. | through study completion, an average of 4 years
  Feasibility outcome. The term 'withdrawal' encompasses two potential scenarios; withdrawal due to loss of consent or withdrawal due to death.
Quality of life and resource data collection - Sf12. | through study completion, an average of 4 years
  Feasibility outcome. Feasibility of quality of life and resource data collection will be assessed for data completeness and consistency using Sf12.
Quality of life and resource data collection - EQ5D. | through study completion, an average of 4 years
  Feasibility outcome. Feasibility of quality of life and resource data collection will be assessed for data completeness and consistency using EQ5D.
Quality of life and resource data collection - HADS. | through study completion, an average of 4 years
  Feasibility outcome. Feasibility of quality of life and resource data collection will be assessed for data completeness and consistency using HADS.
Quality of life and resource data collection - VAS. | through study completion, an average of 4 years
  Feasibility outcome. Feasibility of quality of life and resource data collection will be assessed for data completeness and consistency using VAS.
Quality of life and resource data collection - patient diary. | through study completion, an average of 4 years
  Feasibility outcome. Feasibility of quality of life and resource data collection will be assessed for data completeness and consistency using patient diary.

SECONDARY OUTCOMES:
Days with immobilisation | through study completion, an average of 4 years
  Days with immobilisation measured at the end study.
Progression of foot deformity as documented by measuring radiological foot alignment angles. | Six months after remission.
  All x-rays will be taken in a weight bearing position with standard views as per WPD. Comparison from baseline, diagnosis of remission, and six months after remission.

OTHER OUTCOMES:
Pain in the foot, ankle or leg measured, using the Numeric Pain Rating Scale. | At randomisation, and three monthly until patient is in remission. Also collected at 1 month and 6 months post remission
  Patient Reported Outcome Measures - VAS - Visual Analogue Scale. Minimum value 0 (no pain at all) Maximum 100 (pain as bad as it could possibly be)
Health related quality of life. | At randomisation, and three monthly until patient is in remission. Also collected at 1 month and 6 months post remission
  Patient Reported Outcome Measures. Health related quality of life assessed by the Medical Outcomes Short-Form Health Questionnaire (SF12) - Sf12 - Short form 12 health related quality of life questionnaire. Not a scale.
Psychological health status. | At randomisation, and three monthly until patient is in remission. Also collected at 1 month and 6 months post remission
  Patient Reported Outcome Measures. Psychological health status measured using the Hospital Anxiety and Depression Scale (HADs) - HADS - Hospital Anxiety and Depression Scale. Participant selects statements that best reflect their feelings. Not a numbered scale.
EQ-5D-5L | At randomisation, and three monthly until patient is in remission. Also collected at 1 month and 6 months post remission
  Patient Reported Outcome Measures - EQ-5D-5L - health related quality of life questions across five dimensions. One scale used for participant to reflect how they feel their health is on the day of completion. Scale is 0-100, 0 is the worst health imaginable and 100 is the best health imaginable
Economic Evaluation - Reported through a patient diary | At randomisation, and three monthly until patient is in remission. Also collected at 1 month and 6 months post remission
  Patient Reported Outcome Measures. Collecting resource use and quality of life data, to inform the design of the health economics component of a future definitive trial - Participant asked if working and if this has changed because of their condition. Also asked to indicate if there are any costs associated with attendance at medical appointments (travel and/or parking).

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Gooday, Study Chair — Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK)
Locations (1):
- Norfolk & Norwich University Hospital, Norwich, Norfolk, United Kingdom

DOCUMENTS (1):
  • Study Protocol (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT05104944/Prot_000.pdf